CLINICAL TRIAL: NCT04826237
Title: Towards a Self-Administered Hearing Protection Regimen
Brief Title: Oral Statins and Protection From Hearing Loss
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Donna S Whitlon, Research Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STU00212929
Record Dates: First submitted 2021-02-24; First posted 2021-04-01 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Sudden Sensorineural Hearing Loss
Keywords: deafness; statin; hearing loss
MeSH Terms: conditions — Hearing Loss, Sudden; Deafness; Hearing Loss | interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors; Methylprednisolone; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Neither the participant, the medical professionals, nor those that initially calculate the testing data will know which patient has the placebo or which has the statin. Each patient will be identified by number and sex. Only the clinical coordinator who records the names and treatments and the principal investigator (who does not see patients) will have access to the key. The drugs will be randomized in two groups (for female and male). No one doing data analysis will have any identifiable information other than sex and when the code is broken, the data will be tagged with the identification number of hte patient
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Statin (Experimental): Methylprednisolone+statin (identity and dose to be determined before Trial Begins) Oral methyprednisolone, tapering dose over 11 days, beginning at 16 mg 4 x a day;
  Oral statin 1 dose per day for 7 days, beginning with the first dose of methylprednisolone:
  If no improvement after two weeks, offer up to 2 doses intratympanic dexamethasone (10 mg/cc) 10 days apart.
  Interventions: Drug: Statin; Drug: methylprednisolone; Drug: dexamethasone
- Placebo (Placebo Comparator): Methylprednisolone+ placebo. Oral methyprednisolone, tapering dose over 11 days, beginning at 16 mg 4 x a day; Oral placebo 1 dose per day for 7 days, beginning with the first dose of methylprednisolone
  If no improvement after two weeks, offer up to 2 doses intratympanic dexamethasone (10 mg/cc) 10 days apart.
  Interventions: Drug: methylprednisolone; Drug: dexamethasone; Drug: Placebo

INTERVENTIONS:
Drug: Statin — Oral dose to be taken with methylprednisolone
  Other Names: HMG-coA reductase Inhibitor
  Arms: Statin
Drug: methylprednisolone — oral dose, standard of care
  Other Names: medrol
Drug: dexamethasone — Drug for intratympanic administration
  Other Names: decadron
Drug: Placebo — Capsule the same as for statins but without statin
  Arms: Placebo

SUMMARY:
A small clinical trial for idiopathic sudden sensorineural hearing loss (ISSNHL). Will the addition of an oral statin to the standard treatment (oral methylprednesolone and the salvage therapy of intratympanic dexamethasone) improve the treatment outcome for patients with ISSNHL? This study will compare the two treatments and quantitatively evaluate hearing and speech discrimination and have the patients subjectively evaluate tinnitus.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients diagnosed with idopathic sudden sensorineural hearing loss who do not meet the exclusion criteria and do meet the inclusion criteria, and who give written informed consent will be enrolled in the trial. A standard treatment for ISSNHL (oral methyprednisolone) will be given to half of the patients and the other half of the patients will receive the standard treatment plus either a placebo or a 7-day course of an HMG-CoA reductase inhibitor (a statin). Patients will return for follow up, the timing and further treatment of which will be determined by the response to the drugs. At each appointment, the patients will see the medical professional, have a hearing test, a speech in noise test, and self evaluate for tinnitus. If there is no improvement after 2 weeks, patient will be offered up to two intratympanic doses of dexamethasone, 10 days apart. This is a randomized, double-blind prospective study. Randomization of males will be separate from that of females.

ELIGIBILITY:
Inclusion Criteria:

* Patient older than 18 years and younger than 81 years and
* Diagnosed with one sided idiopathic sudden sensorineural hearing loss by physical examination, history, audiology, speech interpretation tests and tinnitus evaluation and
* Seen in the clinic within the first 14 days after the onset of symptoms. and
* Mean hearing threshold equal to or worse than >30 dB averaged across three consecutive frequencies.
* Excellent English Speaking and Comprehension

Exclusion Criteria:

* Children
* Prisoners
* Pregnant women
* Patients who have experienced similar prior events of SSNHL
* Patients with bacterial infections, mycoplasma, Lyme disease, tuberculosis, syphilis, fungal infections,
* Autoimmune inner ear disease
* Middle ear inflammation or effusion
* Ototoxic medication such as chemotherapy, loop diuretics, high dose aspirin, etc.
* Head Trauma, lead poisoning
* Genetic disorders affecting hearing
* Mitochondrial disorders, including MELAS (metabolic encephalopathy, lactic acidosis, and stroke-like episodes), stroke, Cogan's syndrome
* Neoplastic (neurofibromatosis II, bilateral vestibular schwannomas, carcinomatous meningitis, intravascular lymphomatosis, others)
* Sarcoidosis
* Hyperviscosity syndrome
* Diabetes
* Use of statins within the last 12 months
* Allergy, hypersensitivity or intolerance to any components of the study medication
* Prior tinnitus
* Prior otologic surgery other than ventilation tubes
* History of drug abuse or alcoholism within the prior 2 years
* Any psychiatric syndrome requiring treatment with neuroleptics, antidepressants, hypnotics or anxiolytics
* Severe systemic neurologic disease (epilepsy, Parkinson's, dementia/Alzheimers, multiple sclerosis
* Oral steroid treatment within the preceding 30 days
* Heart disease or TIAs
* Chronic kidney failure
* HIV, Hepatitis B or C
* Active shingles
* Skull, facial or temporal bone anomalies

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-02-09 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Pure Tone Audiometry for Hearing Assessment | At the initiation and the end of the study (up to 4 months after initial assessment)
  Pure tone audiometry to calculate Pure tone averages (PTA) at 500 Hz, 1 kHz, 2 kHZ and 4 kHz. will be measured before and at the end of the study. PTA within 15 dB of the pretreatment PTA of the contralateral cochlea will be considered complete improvement.
  At the end of the study, PTA improvement will be compared between experimental and placebo groups, with a difference of 15 dB or more considered a change in response.
  PTA at the end of the study will also be compared between a) males and female groups; b)compared between those presenting for treatment within 1 week of loss of hearing and those presenting between 1 week and 2 weeks; c) PTA will also be determined and compared between different age groups.
  PTA at the end of the study together with word recognition scores at the end of the study will be used to determine the class of hearing improvement using the Gardner-Robertson Scale.
Change in Speech Discrimination | At the initiation and the end of the study, up to 4 months after initial assessment
  At the beginning and the end of the study, word recognition improvement will be compared a) between experimental and placebo groups;b) between males and female groups; c) compared between those presenting for treatment within 1 week of loss of hearing and those presenting between 1 week and 2 weeks; d) word recognition scores will also be and compared between different age groups.
  At the end of the study, Word recognition score (% correct). will be used with the PTA at the end of the study to to calculate the Gardner-Robertson classification of hearing improvement.
Change in Tinnitus Score | AT the initiation and the end of the study, up to 4 months after initial assessment
  Tinnitus Handicap Index; A 6 point or better change in the index indicates improvement.
  AT the end of the study, Tinnitus Index improvement (change) will be compared a) between experimental and placebo groups; b) between males and female groups c); compared between those presenting for treatment within 1 week of loss of hearing and those presenting between 1 week and 2 weeks; and d)

CONTACTS AND LOCATIONS:
Overall Officials: Donna Whitlon, Ph.D., Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
Only unidentified data will be shared